CLINICAL TRIAL: NCT03660566
Title: Use of Leucocyte- and Platelet-rich Fibrin (L-PRF) Membranes in Single Implant Placement on Esthetic Area. Randomized Clinical Trial
Brief Title: Use of Leucocyte- and Platelet-rich Fibrin Membranes in Single Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Maria Aparecida Neves Jardini, Clinical Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Implante PRF
Record Dates: First submitted 2018-07-04; First posted 2018-09-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Tooth Loss; Recession, Gingival
Keywords: Platelet-Rich Fibrin; Dental Implant
MeSH Terms: conditions — Tooth Loss; Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - Implant with L-PRF (Experimental): Patients requiring single implants placement in the esthetic area of maxilla will receive the implant placement with the use of Leucocyte- and Platelet-rich fibrin (L-PRF) membranes.
  Interventions: Procedure: Test - Implant with L-PRF
- Control - Implant without L-PRF (Active Comparator): Patients requiring single implants placement in the esthetic area of maxilla will receive the implant placement only.
  Interventions: Procedure: Control - Implant without L-PRF

INTERVENTIONS:
Procedure: Test - Implant with L-PRF — The patient's blood will be collected and the tubes (4) will be inserted into a tabletop centrifuge (Kasvi). Using a 2500rpm for 12 minutes protocol, the leucocyte- and platelet-rich fibrin clot will be prepared using a kit consisting of a perforated metal box where the clots will be positioned and covered by a metal plaque. The pressure exerted on the clot will lead to the formation of L-PRF membranes, which will be used to cover the ridge after placement of the implant. Then, the flap will be sutured.
  Other Names: Single implant placement with the use of L-PRF membranes
  Arms: Test - Implant with L-PRF
Procedure: Control - Implant without L-PRF — Single implant installation surgery in maxillary esthetic area.
  Other Names: Single implant placement without the use of L-PRF membranes
  Arms: Control - Implant without L-PRF

SUMMARY:
The objective of this randomized controlled clinical trial is to evaluate the increase of soft tissue thickness around single implants installed in maxillary esthetic area with the use of Leucocyte-Platelet rich Fibrin (L-PRF) membranes. The sample is of 42 individuals, where the control group (n = 21) will receive single implant placement only, while the test group will receive single implant placement with L-PRF membranes.

DETAILED DESCRIPTION:
The greatest challenge in implantology is to achieve a satisfactory esthetic result. A new platelet concentrate protocol, named Leucocyte and platelet-rich Fibrin (L-PRF), has been developed in France. Research has shown positive results using L-PRF during implant placement, as improving soft tissue healing and bone formation, leading to higher esthetic level and greater implant stability. The aim of this study is to evaluate if the use of PRF associated to implant placement in esthetic area presents superior aesthetic result and soft tissue thickness increase when compared to implant placement without graft. Forty-two patients requiring single implant placement in the esthetic area of the maxilla will be randomly divided into test group (implant + L-PRF) and control group (implant without graft). Surgical procedures will be performed by a single operator. The rates of soft tissue thickness, esthetic and comfort will be evaluated at baseline and 3 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 20 years of age, systemically healthy, with satisfactory oral hygiene assessed by plaque index and gingival index of less than 25% (O'Leay et al. 1972).
* Patients requiring single implant placement in anterior maxilla (premolar to premolar)
* Buccal soft tissue thickness of at least 2mm
* Patients who agreed to participate in the study and signed a written consent (Resolution nº196 of October 1996 and the Code of Professional Ethics Dental - C.F.O. - 179/93)

Exclusion Criteria:

* Smokers
* Patients with parafunctional habits, such as bruxism
* Patients who need other types of rehabilitation, such as removable prostheses
* Pregnant or lactating
* Patients with uncontrolled systemic diseases (cardiovascular alterations, blood disorders, diseases that affect bone metabolism, immunodeficiencies, diabetes)
* Patients who use drugs that interfere with wound healing or contraindicate the surgical procedure, such as gingival growth related drugs
* Implants in adjacent regions
* Sites requiring bone augmentation procedure
* Patients in orthodontic treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Gain of peri-implant soft tissue thickness | Three months
  A single investigator, who is not the operator, is responsible for the measurements of the patients. The examiner will be judged calibrated. The calibration will be made by examination of soft tissue thickness of 5 patients, twice, in a range of 48 hours. The correlation test will be used to verify the reproducibility of intra-examining measures, with a maximum value of 0.8. To ensure that the measures at baseline and postoperative evaluation will be performed at the same place, we will use a stent, made of condensation silicone (Optosil - Heraeus Kulzer), so as to cover the edentulous region and the regions of interest described by Zeltner et al. (2017). During measurements of soft tissue thickness, the stent will be used so that the tissue perforation site will be standardized, according to a marking on its surface. An endodontic spacer will be used for tissue perforation, and the thickness will be evaluated using a digital caliper.

SECONDARY OUTCOMES:
a) Plaque index (IP, Ainamo e Bay. 1975) | Three months
  Assessment of presence or absence of plaque in a dichotomous pattern (0 - absence of visible plaque; 1 - presence of visible plaque);
b) Gingival bleeding index (IG, Ainamo & Bay, 1975) | Three months
  Assessment of presence or absence of bleeding in the gingival margin in a dichotomous pattern (0 - no bleeding; 1 - presence of bleeding)
c) Buccal keratinized tissue thickness (ETQv) | Three months
  Keratinized tissue thickness measured at the center of the region of interest (RDI) of the buccal surface of the ridge. To measure the tissue thickness, a guiding device will be made to standardize the region to be measured and then, at a specific point, the mucosa will be punctured with an endodontic spacer and the thickness marked with a rubber marker. Then, using a digital caliper, the thickness will be measured.
d) Ridge defect (DR) (ridge valley) | Three months
  Distance in millimeters from the buccal mucosa to the imaginary line passing through the vestibular bosses of the adjacent teeth, using a periodontal probe.
e) Soft tissue height (ATM) | Three months
  Distance from the top of the gingival tissue on the edge of the ridge to the top of the stent, measured using a endodontic spacer with rubber marker to measure height, and then measure with a digital caliper.
f) Height of keratinized tissue (ATQ) | Three months
  Vertical distance in millimeters measured on the center of the ridge on the buccal aspect of the edentulous ridge to the mucogingival line, using a periodontal probe.
g) Distance between the teeth adjacent to the edentulous space (DED) | Three months
  Measure of the distance between the proximal faces of the teeth adjacent to the edentulous area, using a periodontal probe.
h) Vestibular bone plate thickness (ETV) | During the surgical procedure
  The thickness of the buccal bone plate, measured in millimeters, after the perforations of the ridge prior to implant installation. Measured using photos taken during the surgery.
i) Distance between implant and adjacent teeth (DEID) | During the surgical procedure
  Measurements between the implant to the adjacent teeth, mesial and distal. measured using photos taken during the surgery.
j) Distance from the implant to the imaginary line passing by the buccal aspect of the adjacent teeth (DILIV) | During the surgical procedure
  Measured from the vestibular aspect of the implant to the imaginary line passing through the buccal faces of the adjacent teeth. Measured using photos taken during the surgery.
k) Distance from the buccal bone plate to the imaginary line of the adjacent teeth (DTOVLI) | During the surgical procedure
  Measured from the buccal bone plate to the imaginary line of the buccal faces of the adjacent teeth, measured using photos taken during the surgery.
l) Distance from the interproximal bone crest to the cementum-enamel junction of neighboring teeth (DCOJCE) | During the surgical procedure
  Linear measurement from the top of the bone crest to the JCE of the mesial and distal neighboring teeth to the edentulous space (with a periodontal probe)
m) Evaluation of the periodontal biotype (thin or thick) | Three months
  Classified on thin or thick periodontal biotype, according to Olsson and Lindhe, 1991 and Kan et al., 2010. Thin, if the marginal vestibular gingiva is more delicate, the papillae are high and thin and the crown of the central incisors are triangular shaped; Thick if the marginal gingiva is thicker, papillae are short and the central incisors are square shaped.

OTHER OUTCOMES:
Aesthetic (based on the patient's opinion) | One year
  With a hand mirror, the patient will evaluate peri-implant aesthetic immediately after the installation of the final crown and will be asked to mark, on a Visual Analogic scale (VAS), where the left end of the scale will be "very ugly" and the right "very beautiful ". The right end is the best outcome possible.
Postoperative discomfort | Seven days
  After the implant installation, the patients will be asked to mark, on a Analogic Visual scale (VAS), the postoperative discomfort, where the scale results are "none" in the left and "extreme", in the right. The right end is the best outcome possible.
Postoperative discomfort (based on analgesics) | Seven days
  Patients will be asked to report the number of analgesics ingested on a week. Patients should fill out a chart during the first 7 days after the surgery, at home.
  The best result will be if patients do not take analgesics, or ingested as little as possible, which would show that there was no postoperative pain.
Evaluation of oral health impact on quality of life, using the Oral Health Impact Profile (OHIP-14) questionnaire. | One year
  Evaluate the impact of oral health on patient's quality of life before and 1 year after implant installation. This evaluation will be carried out through the application of a questionnaire with 14 questions (Oral Health Impact Profile: OHIP-14) that assess the patient's perception regarding the impact of oral conditions on their well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Jardini, Doctor, Principal Investigator — State of São paulo University
Locations (1):
- Maria Jardini, São Jose Dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No